CLINICAL TRIAL: NCT00235417
Title: Stem Cell Therapy in Chronic Ischemic Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Stem cell
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Last update posted 2007-06-08 (Estimated); Status verified 2007-06

CONDITIONS: Myocardial Ischemia; Heart Failure, Congestive
Keywords: Bone Marrow Transplantation
MeSH Terms: conditions — Myocardial Ischemia; Heart Failure | interventions — Bone Marrow Transplantation

INTERVENTIONS:
Procedure: Bone marrow transplantation

SUMMARY:
The purpose of this study is to determine whether intracoronary bone marrow transplantation can improve left ventricular ejection fraction in patients with severe ischemic heart failure and no other option for standard therapies (revascularization and drugs).

DETAILED DESCRIPTION:
Despite standard therapies (revascularization and drugs), patients with severe ischemic heart failure have a high morbidity and mortality.

The purpose of this study is to determine whether intracoronary transfer of autologous bone marrow cells can induce angiogenesis, subsequently improving regional myocardial perfusion, and finally resulting in improved systolic and diastolic left ventricular function in patients with severe ischemic heart failure.

35 patients with stable left ventricle function will - with four months interval - receive two treatments with bone marrow transplantation intracoronary in vessels supplying dysfunctional myocardial territories. Echocardiography is performed three times prior (four and two months and just before) and two times after (four and eight months after) therapy. It is a non-randomised trial, patients will enter as their own control.

ELIGIBILITY:
Inclusion Criteria:

1. Severe ischemic heart failure and no other other option for standard therapies (revascularization and drugs),
2. Stable left ventricular ejection fraction < 40%,
3. CCS class 2-3 and/or NYHA class 2-3, and
4. Signed informed consent.

Exclusion Criteria:

1. Implantation of pacemaker (including implantable cardioverter defibrillator [ICD] and biventricular pacing),
2. Acute myocardial infarction within 3 months,
3. Atrial fibrillation, or
4. Severe comorbidity that could impact the patient's short-term survival (including primary hematologic disorders)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2005-10; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Changes in left ventricular ejection fraction from baseline to 12 months' follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Per Thayssen, MDSci, Study Director — Department of Cardiology, Odense University Hospital; Axel CP Diederichsen, phd, Principal Investigator — Department of Cardiology, Odense University Hospital
Locations (1):
- Department of Cardiology, Odense University Hospital, Odense, Odense C, Denmark

REFERENCES:
- [Derived] Diederichsen AC, Moller JE, Thayssen P, Videbaek L, Saekmose SG, Barington T, Kassem M. Changes in left ventricular filling patterns after repeated injection of autologous bone marrow cells in heart failure patients. Scand Cardiovasc J. 2010 Jun;44(3):139-45. doi: 10.3109/14017430903556294. PMID 20233136